CLINICAL TRIAL: NCT00592943
Title: A PET Study Examining the Dopaminergic Activity of Armodafinil in Adults
Brief Title: PET Study Examining the Dopaminergic Activity of Armodafinil in Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Thomas J. Spencer, MD, Associate Chief, Clinical and Research Program, Pediatric Psychopharmacology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2007-P-001659
Record Dates: First submitted 2007-12-28; First posted 2008-01-14 (Estimated); Results first posted 2011-06-10 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
Keywords: Adults; Healthy Volunteers; Nuvigil; Armodafinil; DAT occupancy in healthy volunteers
MeSH Terms: interventions — Modafinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Armodafinil (100mg) (Active Comparator)
  Interventions: Drug: armodafinil
- Armodafinil (250 mg) (Active Comparator)
  Interventions: Drug: armodafinil

INTERVENTIONS:
Drug: armodafinil — tablet, taken by mouth, once each study day
  Other Names: Nuvigil

SUMMARY:
The specific aims of this study are 1) to document the Dopamine Transporter (DAT) receptor occupancy of armodafinil using positron emission tomography (PET) scanning with C-11 altropane as the ligand and 2) to document the increased intrasynaptic dopamine produced by armodafinil using PET scanning with C-11 raclopride as the ligand. We hypothesize that DAT occupancy will be low with armodafinil; less than the DAT occupancy produced by therapeutic doses of methylphenidate. We also hypothesize that increases in intrasynaptic dopamine will be relatively low with armodafinil.

DETAILED DESCRIPTION:
Modafinil produces a unique spectrum of pharmacological effects including enhanced vigilance, arousal, and wakefulness in human subjects (Bastuji and Jouvet 1988). The drug is widely used to treat narcolepsy (Banerjee, Vitiello et al. 2004), but is also effective in Attention Deficit Hyperactivity Disorder (ADHD) (Biederman, Swanson et al. 2005). Notwithstanding the expanding clinical indications for modafinil, the neurochemical mechanisms that produce therapeutic improvement remain unresolved. Pre-clinically, modafinil is a weak inhibitor of the DAT, and displays no affinity for dopamine receptor subtypes (Mignot, Nishino et al. 1994). Further evidence supporting low dopaminergic activity is the low abuse potential of modafinil (Jasinski 2000). Various theories have been proposed as alternative modes of action including enhancement of glutamate release and inhibition of Gamma-aminobutyric acid (GABA) release in various brain regions (Ferraro, Antonelli et al. 1997; Ferraro, Antonelli et al. 1997; Ferraro, Antonelli et al. 1999). However, the exact mechanisms of action of modafinil and the principle active metabolite, armodafinil, are unknown. Understanding these mechanisms of action is important in assessing the potential therapeutic role of armodafinil. We will test to see if there are differences in the degree of DAT occupancy and D2 binding of armodafinil compared with that of traditional stimulants.

The main target of typical stimulants in the brain is the dopamine transporter (DAT) (Volkow, Wang et al. 1998). We have an exquisitely sensitive methodology to measure DAT occupancy using C-11 altropane and Positron Emission Tomography (PET) (Fischman, Bonab et al. 2001). Our group has previously documented the central nervous system pharmacokinetics of several psychiatric drugs (including methylphenidate) using similar techniques. (Christian, Livni et al. 1996; Fischman, Bonab et al. 1996; Fischman, Alpert et al. 1997; Salazar and Fischman 1999; Fischman, Alpert et al. 2002; Spencer, Biederman et al. 2006).

Increases in intrasynaptic (extracellular) dopamine concentrations associated with medications are routinely measured by changes in C-11 raclopride binding in PET scans. C-11 raclopride binds to postsynaptic D-2 receptors. If the intrasynaptic concentration of dopamine increases, it competes with raclopride leading to a weaker signal (i.e. decreased raclopride binding to D-2 receptors). After administration of a stimulant, associated increases in intrasynaptic dopamine compete with C-11 raclopride binding in this manner (Volkow, Wang et al. 2002). By using this technology we can document the change in D-2 binding in the intrasynaptic space achieved by armodafinil, and compare it to that achieved by a typical stimulant.

To this end, using two PET ligands (C-11 altropane and C-11 raclopride), this protocol seeks to compare the DAT receptor occupancy and the increased intrasynaptic dopamine produced by armodafinil to previous studies of methylphenidate. This research will provide novel and unique information toward better understanding the mechanisms of action of armodafinil in comparison to those of typical stimulants.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent to participate in the study.
2. Age: 18 - 35
3. If female, non-pregnant, non-nursing with a negative serum pregnancy test and using an adequate form of birth control.
4. Supine and standing blood pressure within the range 110/60 to 150/95 mmHg.
5. Heart rate, after resting for 5 minutes, within the range 46-90 beats/min.
6. Right-handed.

Exclusion Criteria:

1. Diagnosis of any psychotic disorder, bipolar disorder, severe depression, severe anxiety, or Autism.

   Subjects with mild mood, oppositional, conduct, and anxiety disorders may be permitted to participate if considered appropriate by the investigator.
2. Scores of Baseline Scales:

   Hamilton Depression Scale > 17 (out of a possible 67 on the 21-item scale)(Hamilton 1960) Beck Depression Inventory > 19 (out of a possible 63 on the 21-item scale)(Beck, Ward et al. 1961) Hamilton Anxiety Scale > 21 (out of a possible 56 on the 14-item scale) (Hamilton 1959)
3. Tics or Tourette's Syndrome.
4. History of head trauma with loss of consciousness, organic brain disorders, seizures, or neurosurgical intervention.
5. Any clinically significant chronic medical condition, in the judgment of the investigator.
6. Mental impairment as evidenced by an I.Q. <75.
7. Exposure to dopamine receptor antagonists within the previous three (3) months.
8. Exposure to radiopharmaceuticals within four (4) weeks prior to PET scan.
9. Subjects receiving psychotropic medication.
10. Any clinically significant abnormality in the screening laboratory tests, vital signs, or 11-lead ECG, outside of normal limits.
11. Any woman of childbearing potential who is seeking to become pregnant or suspects that she may be pregnant.
12. Subjects with a known recent history (within the past six (6) months) of illicit drug or alcohol dependence.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2007-10; Primary Completion 2008-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Spencer, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States

REFERENCES:
- [Derived] Spencer TJ, Madras BK, Bonab AA, Dougherty DD, Clarke A, Mirto T, Martin J, Fischman AJ. A positron emission tomography study examining the dopaminergic activity of armodafinil in adults using [(1)(1)C]altropane and [(1)(1)C]raclopride. Biol Psychiatry. 2010 Nov 15;68(10):964-70. doi: 10.1016/j.biopsych.2010.08.026. PMID 21035624
- See also: Related Info — http://massgeneral.org/pediatricpsych/home.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twelve healthy human subjects between 18 and 55 years old were sequentially recruited from advertisements.
Pre-assignment Details: 12 healthy human subjects were enrolled and completed the study. Enrollment was gender-balanced. Six subjects (3 males, 3 females) were be randomly assigned to the C-11 altropane group; six subjects (3 males, 3 females) were be randomly assigned to the C-11 raclopride group, all in an open-label protocol.
Groups:
- Armodafinil (100mg): One 100 mg orally administered dose of Armodafini before PET scan.
- Armodafinil (250mg): One 250 mg orally administered dose of Armodafini before PET scan.
Period: Overall Study
Arm/Group | Armodafinil (100mg) | Armodafinil (250mg)
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Armodafinil (100mg) | Armodafinil (250mg) | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Full Range); unit: Years] | 25.13 (1.1) [22.83 to 34.5] | 21.44 (2.5) [18.75 to 22.92] | 23.29 [18.75 to 34.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Armodafinil DAT Occupancy in Caudate
Description: Subjects received each dose level (100 and 250 mg) of armodafinil, followed by PET scans, in an open-label protocol. Repeat PET scans, using [1 1 C]altropane, determined DAT occupancy at 1 hour and 2.5 hours postdose (compared with baseline).
Time Frame: DAT occupancy was measured using the PET scan at 1 hour and 2.5 hours after oral administration of 100mg or 250 mg Armodafinil
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Armodafinil (100mg) | Armodafinil (250mg)
Number analyzed (Participants) | 6 | 6
μg/mL
  1 Hour | 34.0 (9.0) | 60.5 (7.4)
  2.5 hours | 40.4 (9.5) | 65.2 (6.1)

2. Primary Outcome: Armodafinil Extracellular Dopamine in Caudate at 2.5 Hours (With Outlier)
Description: Each subject received each dose level (one dose per day of 100 or 250 mg) of armodafinil, followed by PET scans using [11C]raclopride, to determine the change in extracellular dopamine at 2.5 hours postdose.
Time Frame: Extracellular DAT was measured using the PET scan at 2.5 hours after oral administration of 100mg or 250 mg Armodafinil on three different study visits
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Armodafinil (100mg) | Armodafinil (250mg)
Number analyzed (Participants) | 6 | 6
μg/mL | 17.8 (30.1) | 7.0 (8.6)

3. Primary Outcome: Armodafinil Extracellular Dopamine in Caudate at 2.5 Hours (Without Outlier)
Description: as for outcome 2
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Armodafinil (100mg) | Armodafinil (250mg)
Number analyzed (Participants) | 5 | 5
μg/mL | 6.0 (9.4) | 5.3 (8.5)

ADVERSE EVENTS:
Arm/Group | Armodafinil (100mg) | Armodafinil (250mg)
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/6 | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Armodafinil (100mg) (N=6) | Armodafinil (250mg) (N=6)
slightly jittery (Nervous system disorders) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 1 (2) | 1 (2)
cold/ congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
muscle soreness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 0 (0) | 1 (1)
hyperactivity (Nervous system disorders) | 0 (0) | 1 (1)
shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Extracellular dopamine could compete with [11C] altropane, causing an overestimation of DAT occupancy. Time between scans and menstrual cycle could be sources of variability. Brain pathology although unlikely in normal subjects, is possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No